CLINICAL TRIAL: NCT05893706
Title: The Effect of Single Task vs. Dual Task Assessment on Muscle Strength and Performance in Individuals With Knee Osteoarthritis
Brief Title: The Effect of Single Task vs. Dual Task Assessment in Individuals With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: E-10840098-772.02-3002
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Osteo Arthritis Knee
Keywords: dual task

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dual task: A dual-task paradigm is a procedure in experimental neuropsychology that requires an individual to perform two tasks simultaneously, in order to compare performance with single-task conditions.
- Single task: Single task

SUMMARY:
Osteoarthritis is characterized by progressive degeneration of articular cartilage, weakening of subchondral bone, synovial inflammation, meniscal degeneration, and intra-articular osteophytes.

DETAILED DESCRIPTION:
Dual tasking is when two tasks can be done simultaneously. A dual task may involve two different simultaneous motor tasks, or it may include a cognitive task in addition to the motor task. Following the additional task given, there may be a decrease in the performance of the main task or in the performance of both tasks.

Decreased balance control can lead to fall injuries that result in serious physical, psychological and social losses. Before the management of this condition, an effective evaluation of balance control in patients with knee osteoarthritis is required.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40-65
* A diagnosis of knee osteoarthritis in at least one of the knees clinically and radiographically according to the criteria of the American Society of Rheumatology
* Findings consistent with stage II-III osteoarthritis
* Pain is between 2 and 7 according to the visual analog scale.

Exclusion Criteria:

* Acute osteoarthritis in the knee
* Comorbid diseases (advanced osteoporosis, vertigo, neurological diseases, etc.), injuries and surgeries for which exercise is contraindicated
* NSAID and similar disease-modifying drug use (Diaserein, Glucosamine, etc.)
* Having exercised regularly in the last 6 months (more than 1 day per week)
* Having undergone arthroplasty surgery
* Intra-articular injection (hyaluronic acid/steroid) administration in the last 6 months

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A second assessment will be done 48 hours after the initial one. It will be completed as a dual job for the second evaluation. The patient will be given activities involving colors and numbers as part of the dual evaluation, and concurrently, after the isokinetic device has assessed the patient's muscle strength, the 30-second sit-and-stand test will assess the patient's function and balance.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Lower extremity muscle strength | 3 days
  In the measurement of lower extremity muscle strength, Quadriceps and Hamstring muscle strength will be measured with an isokinetic dynamometer (CSMI-Cybex Humac-Norm Testing & Rehabilitation System). The knee extension test will be performed in a sitting position. The test foot will be secured with a Velcro strap by placing it on the dynamometer arm 1 inch above the ankle. The lateral epicondyle of the femur will be used as the anatomical reference with which the axis of the dynamometer is aligned. Two different speeds of maximal reciprocal concentric isokinetic knee extension and flexion; will be measured as slow (60°/s, 5 reps, 10 sec. rest) and fast (180°/s, 15 reps, 10 sec. rest)
30 second sit and stand test | 3 days
  It is a functional evaluation test. It measures the time it takes to sit and stand in a 43-centimeter-high chair with back support but no armrests for 30 seconds. After the "Start" command, the participant must stand up fully, then return to the initial sitting position. The participant will be motivated to complete as many full sit-ups as possible within 30 seconds. The score is the total number of sits in 30 seconds.
Western Ontario and MacMaster | one day
  The Western Ontario and MacMaster (WOMAC) questionnaire consists of a series of questions that assess three primary dimensions of osteoarthritis: pain, stiffness, and physical functionThe most commonly used scoring system for the WOMAC is the Likert scale, which ranges from 0 to 4 or 0 to 5 for each item.The maximum score would be 96 (the sum of the maximum scores from the three subscales).
Visual Analog Scale | one day
  Visual Analogue Scale, pain level, right and left extremities were evaluated separately. In addition, three different measurements were taken as rest, activity and night. For individuals, a value of 0 was "no pain"; A value of 10 was defined as "unbearably severe pain". The point marked by the patient was measured with a tape measure, and the examined value was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol hospital, Istanbul, Istanbul Avrupa Kitasi, Turkey (Türkiye)

REFERENCES:
- [Background] Abdallat R, Sharouf F, Button K, Al-Amri M. Dual-Task Effects on Performance of Gait and Balance in People with Knee Pain: A Systematic Scoping Review. J Clin Med. 2020 May 21;9(5):1554. doi: 10.3390/jcm9051554. PMID 32455597